CLINICAL TRIAL: NCT02460354
Title: Use of Metformin to Treat Patients With Congenital Nephrogenic Diabetes Insipidus (NDI)
Brief Title: Metformin and Congenital Nephrogenic Diabetes Insipidus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of effect in initial subjects
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Larry Greenbaum, MD, PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00077633
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Insipidus
Keywords: Congenital nephrogenic diabetes insipidus
MeSH Terms: conditions — Diabetes Insipidus; Diabetes Insipidus, Nephrogenic | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Subjects with congenital nephrogenic diabetes insipidus (NDI) will receive one metformin 500 mg pill orally
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg pill dispensed once orally
  Other Names: Glumetza; Fortamet; Glucophage; Riomet

SUMMARY:
The purpose of this study is to determine whether metformin can increase urine concentration (osmolality) and decrease the amount of urine in patients with congenital nephrogenic diabetes insipidus (NDI).

DETAILED DESCRIPTION:
Nephrogenic diabetes insipidus (NDI) is a genetic disease. Patients with this disease make large amounts of urine because their kidneys don't hold on to water. The large amount of urine means that patients need to urinate very frequently. They are also at increased risk for dehydration if they don't drink enough. The large amount of urine can sometimes damage their bladders and kidneys. There are some medicines that may help these patients urinate less, but they are not very effective. There is evidence in animal studies that a medication called metformin may help patients with NDI urinate less.

ELIGIBILITY:
Inclusion Criteria:

* Males with a documented mutation in the vasopressin type 2 receptor (V2R)
* Willing to provide consent and/or assent as appropriate
* Capable of providing urine samples as dictated by the protocol

Exclusion Criteria:

* Urinary incontinence
* Subjects who have heart disease, liver disease, diabetes, cancer, or other significant disease other than Nephrogenic Diabetes Insipidus (NDI)
* Subjects with significant renal dysfunction (defined as a calculated glomerular filtration rate (GFR) <80 ml/min/1.73 m^2)
* Subjects with acquired NDI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in mean urine osmolality | Baseline, 7 hours
  Urine osmolality is a measure of urine concentration. Urine osmolality will be measured using a Wescor vapor pressure osmometer. A normal range for urine osmolality is approximately 500-850 mOsm/kg water. Change is the difference in average osmolality from baseline to 7 hours.

SECONDARY OUTCOMES:
Change in mean urine volume | Baseline, 7 hours
  Urine volume is a measure of fluid balance. Change from baseline in average volume of urine collected from baseline to 7 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Greenbaum, MD, PhD, Principal Investigator — Emory University; Titilayo Ilori, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Childen's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University Hospital - Atlanta Clinical and Translational Science Institute (ACTSI), Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia